CLINICAL TRIAL: NCT05424978
Title: Application of Standardized Green Channel Treatment System for Ischemic Stroke in Xi 'an
Acronym: Asgctsis
Status: Recruiting | Type: Observational
Sponsor: Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SYLL-2021-024
Record Dates: First submitted 2022-06-01; First posted 2022-06-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Acute Ischemic Stroke; Thrombolysis; Endovascular Treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standardized green channel treatment methods for stroke — The measures include six measures: timely triage by triage desk nurses; Rapid evaluation by emergency room physician; If stroke is suspected, the green channel for nosocomial stroke should be activated immediately. Stroke greenway doctors and stroke nurses accompanied patients to complete CT examination; Intravenous thrombolysis in emergency rooms or CT rooms; Suspected macrovascular disease, if the onset time is less than 6 hours, quickly go to the catheter room for intravascular treatment; If the onset time was more than 6 hours, multi-mode imaging was used to quickly evaluate the ischemic penumbra and vascular occlusion, and then the patients were sent to the catheter room for intravascular treatment as soon as possible.

SUMMARY:
Objective: To observe the practical application of the standardized green channel treatment system for stroke in Xi 'an in the real world. Methods: Clinical data and information of patients with acute ischemic stroke who received standardized green channel treatment for stroke were collected, and a multicenter observational clinical study was carried out in the real world to evaluate the prognosis, mortality, incidence of asymptomatic and symptomatic cerebral hemorrhage, incidence of pneumonia, and recurrence rate of stroke after 90 days.

DETAILED DESCRIPTION:
The standardized green channel treatment system for acute ischemic stroke includes: Triage nurse triage timely, rapid assessment emergency doctor, suspected stroke the green channel, immediately start in the green channel of stroke accompanied by doctors and nurses stroke patients improve CT examination, intravenous thrombolysis or CT room, emergency room if considering large vascular lesions and the onset time in 6 hours, and rapidly to international for endovascular treatment, if the onset time of more than 6 hours, Rapid evaluation of ischemic penumbra and vascular occlusion by multi-mode imaging. If there are indications for endovascular treatment, go to the cath room for endovascular treatment as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old;
* Consistent with the diagnosis of acute ischemic stroke;
* 24 hours from onset to enrollment;
* Informed consent

Exclusion Criteria:

* Patients who refuse to receive intravenous thrombolysis or intravascular intervention (including intravascular mechanical thrombolysis and arterial thrombolysis);
* Stroke patients caused by brain tumor, brain trauma and blood diseases;
* Those with a history of stroke and sequelae affecting the outcome assessment, namely, mRS 2 points before the onset of this stroke;
* Combined with claudication osteoarthritis rheumatoid arthritis gout arthritis and other limb dysfunction and affect the neurological function examination;
* Patients with severe hepatic and renal insufficiency (Note: Hepatic insufficiency refers to ALT or AST values greater than 2 times the upper normal limit; Renal insufficiency refers to blood creatinine value greater than 2 times the normal upper limit);
* Suffering from other serious life-threatening diseases with an expected survival time of less than 3 months;
* Other diseases that limit neurological function evaluation or affect patient follow-up;
* A woman planning to be pregnant or breastfeeding;
* Currently participating in other clinical trials;
* Refuse to participate in the registration of investigators

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke within 24 hours of onset; Receive standardized green channel treatment for stroke
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of function independent | 90 days after onset
  Rate of modified Rankin Scale(mRS) score less than 3 at 90 days

SECONDARY OUTCOMES:
Rate of mortality | 90 days after onset
  90-day mortality rate
Rate of stroke recurrence | 90 days after onset
  90-day stroke recurrence rate
Rate of cerebral hemorrhage and pneumonia | During hospitalization.
  Incidence of cerebral hemorrhage and pneumonia after thrombolysis or intravascular therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ye Tian, Doctor, Study Director — The dean
Locations (1):
- Xi 'an No.3 Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
Data is managed by the project team and can be shared according to individual needs